CLINICAL TRIAL: NCT04531787
Title: Persistence of Influenza Vaccine-induced Antibodies in Lung Transplant Patients Between Seasons
Brief Title: Influenza Vaccine in Lung Transplant Patients - Persistence of Antibodies
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2004-0240c; A561000 (Other: UW Madison); PHARM/PHARMACY/PHARMACY (Other: UW Madison)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Influenza
Keywords: Pre or post-lung transplant; Healthy
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vaccine, Pre-transplant: cohort consists of individuals waiting for lung transplantation. Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine
- Vaccine, Post-transplant: Cohort consist of individuals who have received lung transplants Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine
- Vaccine, Healthy Controls: Cohort consists of healthy individuals who received the influenza vaccine Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine

INTERVENTIONS:
Drug: Influenza vaccine — influenza vaccine 0.5 ml intramuscularly each season: 2004-2005, 2005-2006, 2006-2007, 2007-2008 for season specific A/H1N1, A/H3N2, and B antigens

SUMMARY:
This a sub-study of a 5-year study designed to investigate how antibody and T cell responses following influenza vaccine compare among lung transplant patients, patients waiting for lung transplantation, and healthy individuals.

This study is designed to investigate influenza vaccine-induced antibodies in lung transplant patients between seasons.

DETAILED DESCRIPTION:
In the recent past, immunization policy-making bodies advised against immunizing too early in the influenza season because vaccine-specific antibody may wane before the end of the influenza season. This recommendation was based on only a small amount of data in frail elderly individuals, and further examination of the evidence shows that influenza vaccine antibody may last much longer. The influenza immunization timing recommendation is now changed to immunize when vaccine is available and continue throughout the season.

These changes led the investigators to the question of duration of influenza vaccine-induced antibody in lung transplant patients. No published studies of antibody persistence in this population could be found.

As part of a 5-year study of influenza antibody response in lung transplant patients, in patients awaiting lung transplantation, and in healthy controls, serum was obtained before and 2-4 weeks after influenza immunization for each season. Therefore, a serum sample was collected on each participant approximately 11 months after influenza vaccine administration for each of 4 years.

To investigate duration of influenza antibody titers, antibody concentrations to the previous season's vaccine antigens were measured.

The hypothesis is that immunosuppressed lung transplant patients would maintain protective concentrations of influenza antigen-specific antibodies (an antibody titer of at least 1:40) beyond the influenza season.

[This substudy that was originally registered to NCT00205270 and subsequently registered to its own NCT number for the purpose of clarity in linked results]

ELIGIBILITY:
Inclusion Criteria:

* Receiving care pre- or post-lung transplant at University of Wisconsin Hospital
* Healthy adult

Exclusion Criteria:

* Allergy to eggs
* Moderate to severe febrile illness
* Active treatment for acute rejection
* Received season's influenza vaccine prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult or patient receiving care pre- or post-lung transplant at University of Wisconsin Hospital
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2004-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Influenza Vaccine Seroprotection at 11 months post immunization | up to 11 months
  A protective influenza antibody concentration is a titer of greater than or equal to 1:40. Influenza antibody concentrations were measured using hemagglutination inhibition assays.

SECONDARY OUTCOMES:
Antibody Concentrations Measured by Geometric Mean Titer | 2-4 weeks post immunization, up to 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Hayney, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moran JJ, Rose WE, Darga AJ, Rohde KA, Hayney MS. Persistence of influenza vaccine-induced antibodies in lung transplant patients between seasons. Transpl Infect Dis. 2011 Oct;13(5):466-70. doi: 10.1111/j.1399-3062.2011.00654.x. Epub 2011 May 27. PMID 21615847